CLINICAL TRIAL: NCT02889666
Title: A Multi-Center and Randomized Control Trial of Cisplatin, Carboplatin, Oxaliplatin, Docetaxel and Gemcitabine Plus Surgery as Treatment for Relapsed and Refractory Non-Small Cell Lung Cancer
Brief Title: A Randomised Trial of Chemotherapy Plus Surgery for Recurrent Non-Small Cell Lung Cancer
Acronym: CCODG-NSCLC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai 10th People's Hospital (Other); Jilin University (Other); Jiangxi Provincial Cancer Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Yu Sun, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCA-81472709
Record Dates: First submitted 2016-08-25; First posted 2016-09-05 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Recurrent Non-small Cell Lung Cancer
Keywords: relapsed; non-small cell lung cancer; cisplatin; carboplatin; oxaliplatin; docetaxel; gemcitabine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence | interventions — Cisplatin; Carboplatin; Docetaxel; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Carboplatin (Experimental): Carboplatin-based chemotherapy (Carboplatin 400mg) was performed 30 days before surgery for patients who had previous surgery to remove the primary non-small cell lung carcinoma but suffered from the recurrent disease. The same chemotherapy using Carboplatin was done for 3 cycles with 30 days after last surgery.
  Interventions: Drug: Carboplatin
- Docetaxel (Experimental): Docetaxel-based chemotherapy (Docetaxel 120mg) was performed 30 days before surgery for patients who had previous surgery to remove the primary non-small cell lung carcinoma but suffered from the recurrent disease. The same chemotherapy using Docetaxel was done for 3 cycles with 30 days after last surgery.
  Interventions: Drug: Docetaxel
- Gemcitabine/Cisplatin (Experimental): Gemcitabine/Cisplatin-based combinational chemotherapy (Gemcitabine 200mg + Cisplatin 60mg) was performed 30 days before surgery for patients who had previous surgery to remove the primary non-small cell lung carcinoma but suffered from the recurrent disease. The same chemotherapy was done for 3 cycles with 30 days after last surgery.
  Interventions: Drug: Gemcitabine/Cisplatin
- Cisplatin (Experimental): Cisplatin-based chemotherapy (Cisplatin 60mg) was performed 30 days before surgery for patients who had previous surgery to remove the primary non-small cell lung carcinoma but suffered from the recurrent disease. The same chemotherapy using Cisplatin was done for 3 cycles with 30 days after last surgery.
  Interventions: Drug: Cisplatin
- Docetaxel/Oxaliplatin (Experimental): Docetaxel/Oxaliplatin-based chemotherapy (Docetaxel 120mg + Oxaliplatin 200mg) was performed 30 days before surgery for patients who had previous surgery to remove the primary non-small cell lung carcinoma but suffered from the recurrent disease. The same chemotherapy was done for 3 cycles with 30 days after last surgery.
  Interventions: Drug: Docetaxel/Oxaliplatin
- Docetaxel/Carboplatin (Experimental): Docetaxel/Carboplatin-based chemotherapy (Docetaxel 120mg + Carboplatin 400mg) was performed 30 days before surgery for patients who had previous surgery to remove the primary non-small cell lung carcinoma but suffered from the recurrent disease. The same chemotherapy was done for 3 cycles with 30 days after last surgery.
  Interventions: Drug: Docetaxel/Carboplatin
- Gemcitabine/Carboplatin (Experimental): Gemcitabine/Carboplatin-based chemotherapy (Gemcitabine 200mg + Carboplatin 400mg) was performed 30 days before surgery for patients who had previous surgery to remove the primary non-small cell lung carcinoma but suffered from the recurrent disease. The same chemotherapy was done for 3 cycles with 30 days after last surgery.
  Interventions: Drug: Gemcitabine/Carboplatin
- Placebo (Placebo Comparator): No Adjuvant chemotherapy using CCODG was done for patients who had previous surgery to remove the primary non-small cell lung carcinoma but subject to tumor relapse. Instead, placebo was supplied to these patients as a comparator Arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cisplatin — Procedure: Preoperative chemotherapy using Cisplatin (60mg) as single agent was performed 30 days before surgery through intravenous (IV) administration. IV administration once every 7 days, totally 4 cycles. There is a 2-day interval between the last dose and surgery.
  Other Names: Platinol
  Arms: Cisplatin
Drug: Carboplatin — Procedure: Preoperative chemotherapy using Carboplatin (400mg) as single agent was performed 30 days before surgery through intravenous (IV) administration. IV administration once every 7 days, totally 4 cycles. There is a 2-day interval between the last dose and surgery.
  Other Names: Paraplatin
  Arms: Carboplatin
Drug: Docetaxel — Procedure: Preoperative chemotherapy using Docetaxel (120mg) as single agent was performed 30 days before surgery through intravenous (IV) administration. IV administration once every 7 days, totally 4 cycles. There is a 2-day interval between the last dose and surgery.
  Other Names: Taxotere
  Arms: Docetaxel
Drug: Gemcitabine/Carboplatin — Procedure: Preoperative chemotherapy using Gemcitabine (200mg) and Carboplatin (400mg) as combinational therapy agent was performed 30 days before surgery through intravenous (IV) administration. IV administration once every 7 days, totally 4 cycles. There is a 2-day interval between the last dose and surgery.
  Other Names: Gemzar/Paraplatin
  Arms: Gemcitabine/Carboplatin
Drug: Gemcitabine/Cisplatin — Procedure: Preoperative chemotherapy using Gemcitabine (200mg) and Cisplatin (60mg) as combinational therapy agent was performed 30 days before surgery through intravenous (IV) administration. IV administration once every 7 days, totally 4 cycles. There is a 2-day interval between the last dose and surgery.
  Other Names: Gemzar/Platinol
  Arms: Gemcitabine/Cisplatin
Drug: Docetaxel/Oxaliplatin — Procedure: Preoperative chemotherapy using Docetaxel (120mg) and Oxaliplatin (200mg) as combinational therapy agent was performed 30 days before surgery through intravenous (IV) administration. IV administration once every 7 days, totally 4 cycles. There is a 2-day interval between the last dose and surgery.
  Other Names: Taxotere/Eloxatin
  Arms: Docetaxel/Oxaliplatin
Drug: Docetaxel/Carboplatin — Procedure: Preoperative chemotherapy using Docetaxel (120mg) and Carboplatin (400mg) as combinational therapy agent was performed 30 days before surgery through intravenous (IV) administration. IV administration once every 7 days, totally 4 cycles. There is a 2-day interval between the last dose and surgery.
  Other Names: Taxotere/Paraplatin
  Arms: Docetaxel/Carboplatin
Drug: Placebo — Regular placebo in replacement of agent-specific chemotherapy was supplied to these patients.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the commonly administered chemotherapeutic agents including cisplatin, carboplatin, oxaliplatin, docetaxel and gemcitabine for solid tumors in clinical oncology, either a single format or given as combinations followed by surgery are effective in the treatment of relapsed and refractory non-small cell lung cancer patients.

DETAILED DESCRIPTION:
Lung carcinoma is a malignant disease characterized by uncontrolled alveolar type II epithelial cell growth in lung tissues. Worldwide in 2012, lung cancer occurred in 1.8 million people and resulted in 1.6 million deaths, making it the most common cause of cancer-related death in men and second most common in women after breast cancer. The most common age at diagnosis is 70 years, and less than 20% of people diagnosed with lung cancer can survive five years post diagnosis. The two main types of lung carcinomas are small cell lung carcinoma (SCLC) and non-small cell lung carcinoma (NSCLC). NSCLC represents the most common type of lung cancers, and approximately 85% of lung cancers are NSCLC. Squamous cell carcinoma, adenocarcinoma, and large cell carcinoma are all subtypes of NSCLC, the latter associated with high mortality in overall cancer populations with limited treatment options.

In this study, the investigators performed a Phase I, open label, agent-combination exploration, multicenter clinical trial to establish the treatment efficacy of several chemotherapeutic agents in patients with recurrent NSCLC who have undergone prior surgery for the primary disease. Up to four cohorts have been enrolled to determine the effectiveness and safety of single or combinational therapeutic strategy. Besides the five-year disease-free survival, overall survival and five-year metastasis-free survival post treatment, the investigators also take into account the anticancer agent-induced tumor stroma damage extent, which may provide further evidence to support the treatment efficacy and assess the potential influence of a damaged tumor microenvironment on disease progression or regression in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 75 years with histologically proven NSCLC
* No severe major organ dysfunction
* WHO performance status of 0 or 1
* No prior cancer chemotherapy
* A Clinical Stage ≥ IA (T1a, N0, M0) of lung disease but without diagnosed distant metastasis (according to the 1997 revision of the International Union Against Cancer TNM staging system) as determined by a preoperative evaluation that included a pleural computed tomography (CT) scan.

Exclusion Criteria:

* Age ≥ 76
* Severe major organ dysfunction
* WHO performance status of >1
* Prior cancer chemotherapy
* Stage IV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-01; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
5 years disease-free survival | 5 years
  The disease-associated survival status during the 5 years post treatment will be measured. Note the information in the Outcome Measure is only study hypothesis.

SECONDARY OUTCOMES:
5 years overall survival | 5 years
  The overall survival status during the 5 years post treatment will be measured. Information in the Outcome Measure is only study hypothesis.
5 years metastasis-free survival | 5 years
  The metastasis-associated survival status during the 5 years post treatment will be measured. Information in the Outcome Measure is only study hypothesis.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Sun, Ph.D, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (3):
- China (3):
  - China-Japan Union Hospital, Jilin University, Changchun, Jilin
  - Shanghai 10th People's Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Tongji University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Yes, there is plan to make individual participant data (IPD) available. According to the medical administration committee of our hospitals, these data will be made generally public upon the completion of the primary studies (anticipated to be July, 2017).